CLINICAL TRIAL: NCT01647659
Title: An Open-Label, Two-Period, Randomized, Crossover Study to Assess the Relative Bioavailability of GSK1120212 Tablet Formulation and the GSK1120212 Pediatric Oral Solution Formulation Following Single-Dose Administration to Adult Subjects With Solid Tumors
Brief Title: Relative Bioavailibilty for Pediatric Powder for Suspension (PfOS) Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 115892
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cancer
Keywords: MEK inhibitor GSK1120212; pharmacokinetics; powder for oral solution; Solid Tumors; pediatric formulation
MeSH Terms: conditions — Neoplasms | interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK1120212 tablet (Experimental): GSK1120212 tablet
  Interventions: Drug: Trametinib tablet
- GSK1120212 powder for oral solution (Experimental): GSK1120212 powder for oral solution
  Interventions: Drug: Trametinib pediatric formulation

INTERVENTIONS:
Drug: Trametinib tablet — 2 mg, orally, on Day 1 of the dosing period
  Arms: GSK1120212 tablet
Drug: Trametinib pediatric formulation — 2 mg, orally, on Day 1 of the dosing period
  Arms: GSK1120212 powder for oral solution

SUMMARY:
The purpose of this open-label, randomized, 2-treatment, 2-period crossover study with incomplete washout is to evaluate the relative bioavailability of 2mg GSK1120212 pediatric oral solution formulation in comparison to 2mg GSK1120212 tablet formulation, to investigate the safety and tolerability of a single dose of the GSK1120212 pediatric oral solution formulation as compared to a single dose of the GSK1120212 tablet formulation, and to investigate the palatability of the GSK1120212 pediatric oral solution formulation.

Subjects will be assigned to one of two possible treatment sequences according to the randomization code provided to the sites by GSK: a single dose of 2mg GSK1120212 pediatric oral solution formulation then a single dose of 2mg GSK1120212 tablet formulation, or a single dose of 2mg GSK1120212 tablet formulation, then a single dose of 2mg GSK1120212 pediatric oral solution formulation. Administration of GSK1120212 in either sequence will be followed by 7 days of serial blood sampling for pharmacokinetic analysis of plasma GSK1120212. Safety assessments, including assessment of adverse events, clinical laboratory values (hematology, clinical chemistry and urinalysis) and vital signs, will be made throughout the study. After completing the pharmacokinetic assessments for two periods, eligible subjects may transition to MEK114375, an open-label rollover study of GSK1120212.

DETAILED DESCRIPTION:
The purpose of this open-label, randomized, 2-treatment, 2-period crossover study with incomplete washout is to evaluate the relative bioavailability of 2mg GSK1120212 pediatric oral solution formulation in comparison to 2mg GSK1120212 tablet formulation, to investigate the safety and tolerability of a single dose of the GSK1120212 pediatric oral solution formulation as compared to a single dose of the GSK1120212 tablet formulation, and to investigate the palatability of the GSK1120212 pediatric oral solution formulation.

Subjects will be assigned to one of two possible treatment sequences according to the randomization code provided to the sites by GSK: a single dose of 2mg GSK1120212 pediatric oral solution formulation then a single dose of 2mg GSK1120212 tablet formulation, or a single dose of 2mg GSK1120212 tablet formulation, then a single dose of 2mg GSK1120212 pediatric oral solution formulation. Administration of GSK1120212 in either sequence will be followed by 7 days of serial blood sampling for pharmacokinetic analysis of plasma GSK1120212. Safety assessments, including assessment of adverse events, clinical laboratory values (hematology, clinical chemistry and urinalysis) and vital signs, will be made throughout the study. After completing the pharmacokinetic assessments for two periods, eligible subjects may transition to MEK114375, an open-label rollover study of GSK1120212.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older, at the time of signing the informed consent.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Able to swallow and retain oral medication.
* Histologically- or cytologically-confirmed diagnosis of a solid tumor malignancy that is not responsive to standard therapies; or for which there is no approved or curative therapy; or for subjects which refuse standard therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate baseline organ function, defined as: absolute neutrophil count >= 1.2X10^9/L; hemoglobin >=9g/dL; platelets >=75X10^9/L; prothrombin time (PT), international normalized ratio (INR) and partial thromboplastin time (PTT) <=1.5 X upper limit of normal (ULN); total bilirubin <=1.5 X ULN; alanine aminotransferase <=2.5 X ULN; creatinine <=1.5 X ULN OR calculated creatinine clearance or 24-hour urine creatinine clearance >= 50mL/min; left ventricular ejection fraction (LVEF) >= lower limit of normal (LLN); systolic blood pressure <140mm Hg
* Women of child-bearing potential must have a negative serum pregnancy test within 14 days of first dose of investigational product administration and agree to use effective contraception, as defined in the protocol, during the study and for 6 weeks following the last dose of investigational product.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until 16 weeks after the last dose of GSK1120212.

Exclusion criteria

* Currently receiving cancer therapy (e.g., chemotherapy with delayed toxicity, extensive radiation therapy, immunotherapy, biologic therapy, or major surgery) within 3 weeks prior to randomization; chemotherapy regimens without delayed toxicity within 2 weeks prior to randomization; or use of an investigational anti-cancer drug within 4 weeks prior to randomization.
* Unresolved Grade 2 or greater toxicity (based on NCI-CTCAE, version 4.0, 2009) from previous anti-cancer therapy except Grade 2 decreased haemoglobin levels or alopecia.
* Pre-existing peripheral neuropathy >= Grade 2.
* Has participated in a clinical trial and received investigational product within 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product, whichever is longer, prior to the first dose of investigational product in this study.
* Has participated in a clinical trial that resulted in or made a donation of blood or blood products in excess of 500mL within 56 days of the first dose of investigational product in this study.
* Has presence of active GI disease or other condition (e.g., gastrectomy, bariatric surgery, small or large bowel resection, or cholecystectomy) that may interfere significantly with absorption of drugs.
* Any serious and/or unstable pre-existing medical (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance with the study procedures, in the opinion of the investigator or the GSK medical monitor.
* History of interstitial lung disease or pneumonitis.
* History or current evidence / risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR), including history of RVO or CSR, or predisposing factors to RVO or CSR (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled systemic disease(s) such as hypertension, diabetes mellitus, or history of hyperviscosity or hypercoagulability syndromes); visible retinal pathology as assessed by ophthalmic exam that is considered a risk factor for RVO or CSR such as evidence of new optic disc cupping, evidence of new visual field defects, or intraocular pressure > 21mm Hg.
* Has symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression; NOTE: Subjects previously treated for these conditions that have had stable central nervous system (CNS) disease (verified with consecutive imaging studies) for >3 months, are asymptomatic and are not currently taking corticosteroids, or are on stable dose of corticosteroids for at least 1 month prior to Day 1 of the study are permitted. Subjects are not permitted to receive enzyme-inducing anti-epileptic drugs (EIAEDs).
* QTcB or QTcF >=480msec.
* Subject has a history or evidence of cardiovascular risk, including any of the following: history or evidence of current clinically significant uncontrolled arrhythmias. Exception: subjects with controlled atrial fibrillation for >30days prior to randomization are eligible OR history of acute coronary syndromes, including myocardial infarction and unstable angina, coronary angioplasty, or stenting, within 6months prior to randomization.
* History or evidence of current >=Class II congestive heart failure as defined by New York Heart Association (NYHA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-07-30 (Actual); Primary Completion 2012-11-12 (Actual); Study Completion 2012-11-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the relative bioavailability of a PfOS formulation relative to the commercial GSK1120212 tablet formulation in adult subjects with solid tumors | 168 hours X 2

SECONDARY OUTCOMES:
Safety and tolerability as determined by the number of patients with adverse events, serious adverse events, and changes in lab values and vital signs from baseline | Day 1 of each dosing session and followup
Evaluate the palatability (bitterness, sweetness, overall taste and aroma) of the pediatric formulation of GSK1120212 | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Nashville, Tennessee

REFERENCES:
- See also: Results for study 115892 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115892?search=study&study_ids=115892#rs